CLINICAL TRIAL: NCT03303053
Title: A Multi-center, Open Label, Randomised Parallel- Group Study to Compare the Efficacy of Cholestyramine Plus Standard Treatment Versus Prednisolone Plus Standard Treatment Versus Standard Treatment Alone in Treatment of Overt Hyperthyroidism
Brief Title: Efficacy and Safety of Cholestyramine and Prednisolone as Adjunctive Therapy in Treatment of Overt Hyperthyroidism
Acronym: ChoPS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChoPS Study Version 3.0
Record Dates: First submitted 2017-09-13; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Hyperthyroidism; Graves Disease
Keywords: Hyperthyroidism,Graves disease,Cholestyramine,Prednisolone
MeSH Terms: conditions — Hyperthyroidism; Graves Disease | interventions — Cholestyramine Resin; Prednisolone; Carbimazole; Propranolol

STUDY DESIGN:
Intervention Model Description: Multi-center, open label, randomised, parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group1:Cholestyramine+standard treatment (Experimental): Cholestyramine powder 4g twice daily, Tablet Carbimazole 30 mg daily, Tablet propanolol 40 mg twice daily for 4 weeks
  Interventions: Drug: Cholestyramine Powder 4g
- Group2:Prednisolone+standard treatment (Experimental): Tablet prednisolone 30 mg daily for week 1, 20 mg daily for week 2, 10 mg daily for week 3 and 5 mg daily for week 4, Tablet carbimazole 30 mg daily, Tablet propanolol 40 mg twice daily for 4 weeks
  Interventions: Drug: Prednisolone
- Group 3: Standard treatment alone (Active Comparator): Carbimazole 30 mg daily and propanolol 40 mg twice daily for 4 weeks
  Interventions: Drug: Standard treatment

INTERVENTIONS:
Drug: Cholestyramine Powder 4g — Cholestyramine powder 4g twice daily, Tablet Carbimazole 30 mg daily, Tablet propanolol 40 mg twice daily for 4 weeks
  Other Names: Questran
  Arms: Group1:Cholestyramine+standard treatment
Drug: Prednisolone — Tablet prednisolone 30 mg daily for week 1, 20 mg daily for week 2, 10 mg daily for week 3 and 5 mg daily for week 4, Tablet carbimazole 30 mg daily, Tablet propanolol 40 mg twice daily for 4 weeks
  Arms: Group2:Prednisolone+standard treatment
Drug: Standard treatment — Carbimazole 30 mg daily and propanolol 40 mg twice daily for 4 weeks
  Other Names: Carbimazole + Propanolol
  Arms: Group 3: Standard treatment alone

SUMMARY:
Hyperthyroidism is the second most common endocrine disorder in the world with Graves' disease being the commonest. Anti thyroid drugs including methimazole, carbimazole, and propylthiouracil are effective treatments but take in most cases between 6 to 8 weeks to achieve euthyroidism. This study aim to assess the efficacy of cholestyramine and prednisolone as adjunctive treatment to standard treatment in patients with overt hyperthyroidism in 4 weeks.

DETAILED DESCRIPTION:
Hyperthyroidism is the second most common endocrine disorder in the world with an estimate prevalence rate of 0.5-1.3% with Graves' disease being the commonest cause.

Uncontrolled hyperthyroidism results in increase cardiovascular morbidity and mortality primarily due to heart failure and thromboembolism. Therefore treatment is essential to restore a euthyroid state in order to reverse the cardiovascular complications.

Anti thyroid drugs (ATDs) including methimazole, carbimazole, and propylthiouracil are effective treatments that inhibit thyroid hormone synthesis, and have clinically important immunosuppressive effects including reducing serum antithyrotropin receptor antibody (TRAb) concentration with time but take in most cases between 6 to 8 weeks to achieve euthyroidism. Therefore there may be a role for adjunctive treatment added on to ATDs. It may be situations where adjunctive treatment is required to alleviate symptoms and restore euthyroidism rapidly such as before surgery or radioactive iodine treatment or in vulnerable groups such as the elderly or those with serious thyrotoxic complications.

This study aim to assess the efficacy of cholestyramine and prednisolone as adjunctive treatment to standard treatment in patients with overt hyperthyroidism in 4 weeks. Cholestyramine is an anion exchange resin that binds thyroxine (T4) in the intestine resulting in fecal excretion of T4 thus reducing the enterohepatic circulation and absorption in hyperthyroidism. Steroids have been shown to be effective in controlling hyperthyroidism by inhibiting the conversion of thyroxine to triiodothyronine peripherally and also blocks the release of thyroxine from the thyroid gland. It may also have the potential to suppress the immune response and hence decrease stimulation of the thyroid gland in Graves.

135 patients with moderate to severe uncontrolled overt hyperthyroid patients secondary to Graves disease will be randomized into 3 groups. Group 1 patients will be treated with cholestyramine 4g twice a day plus carbimazole and propanolol for 4 weeks. Group 2 patients will be treated with prednisolone 30 mg daily for week 1, 20 mg daily for week 2, 10 mg daily for week 3 and 5 mg daily for week 4 plus carbimazole and propanolol for 4 weeks. Group 3 patients will be treated with carbimazole 30 mg daily and propanolol 40 mg bd for 4 weeks. Patients will have their clinical status (weight, blood pressure, pulse rate) measured at baseline along with a TRAb level and Free Triiodotyronine (T3), Free T4 and Thyroid stimulating hormone (TSH) levels. They will be evaluated at week 2 and week 4 of intervention period and have their clinical status (weight, blood pressure, pulse rate) and laboratory (Free T3, Free T4, TSH, Potassium, Fasting/random blood glucose) measured. Adverse events will be monitored at week 2, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written consent by subject or guardian.
2. Subject of either sex, more than 18 years of age
3. Subjects with moderate to severe overt hyperthyroidism (caused by Graves' disease).

   * Moderate to severe overt hyperthyroidism is defined as Free T4> 1.5 times upper limit of normal reference range and TSH below lower limit of reference range, who are either newly diagnosed or previously diagnosed and receiving ATDs currently.
   * Graves disease is defined as hyperthyroidism coupled with clinical signs of symmetrical diffuse goiter, thyroid orbitopathy, or diffuse and vascular thyroid on ultrasound or positive TRAb antibody
4. Female patients will either be

   * post-menopausal for > 2 years
   * Women of childbearing potential can be included if surgically sterile or using double contraception with at least one method being barrier contraception. Women of childbearing potential must have a negative pregnancy test at screening and at randomisation. Pregnancy tests will be repeated during each visit.

Exclusion Criteria:

1. Inability or unwillingness to provide written consent.
2. Inability or unwillingness to comply with the requirements of the protocol as determined by the investigator.
3. Pregnancy, breastfeeding or use of non-reliable method of contraception.
4. Subjects with history of chronic liver disease, chronic renal failure, heart failure, diabetes mellitus
5. Subjects with history of peptic ulcer disease, upper gastrointestinal bleeding, diverticulitis or ulcerative colitis.
6. Subjects who have recently had live or attenuated virus vaccines
7. Subjects with current infection (systemic fungal, active tuberculosis, cerebral malaria, viral hepatitis, HIV)
8. Subjects with cataracts and glaucoma
9. Subjects with osteoporosis
10. Subjects with psychiatric disorders
11. Subjects with complete biliary obstruction, bleeding disorders, hypertriglyceridemia (fasting triglyceride levels > 300mg/dL)
12. Previous history of adverse reactions to cholestyramine or other bile acid sequestrants
13. Previous history of adverse reactions to prednisolone or other steroid compound
14. Current use of cholestyramine or prednisolone or other steroid compound
15. Participation in another clinical trial and/or receipt of cholestyramine or prednisolone within 4 weeks prior to screening visit.
16. Subjects with history of bronchial asthma, bronchospasm, peripheral vascular disease or adverse reactions to propanolol
17. Subjects with adverse reactions to carbimazole
18. Hypokalemia (serum K+ <3.5 mmol/L)
19. Thyroid storm defined as Burch Wartofsky Score >45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients whose Free T4 normalize between the groups | 4 weeks
  Normal Free T4 is defined as Free T4 level between 9-25 pmol/L
Percentage of patients whose Free T3 normalize between the groups | 4 weeks
  Normal free T3 is defined as Free T3 level between 3.5-6.5 pmol/L

SECONDARY OUTCOMES:
Adverse events between the groups | 6 weeks
  Number of adverse events between the groups
Reduction in Free T4 levels | 4 weeks
  Reduction in Free T4 levels ( Change from baseline within 4 weeks)
Reduction in Free T3 levels | 4 weeks
  Reduction in Free T3 levels (Change from baseline within 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Serena SK Khoo, Dr., Principal Investigator — HospitalPutrajaya
Locations (3):
- Malaysia (3):
  - Hospital Putrajaya, Putrajaya, Kuala Lumpur
  - Hospital Queen Elizabeth 2, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nakamura H, Noh JY, Itoh K, Fukata S, Miyauchi A, Hamada N. Comparison of methimazole and propylthiouracil in patients with hyperthyroidism caused by Graves' disease. J Clin Endocrinol Metab. 2007 Jun;92(6):2157-62. doi: 10.1210/jc.2006-2135. Epub 2007 Mar 27. PMID 17389704
- [Background] Hollowell JG, Staehling NW, Flanders WD, Hannon WH, Gunter EW, Spencer CA, Braverman LE. Serum TSH, T(4), and thyroid antibodies in the United States population (1988 to 1994): National Health and Nutrition Examination Survey (NHANES III). J Clin Endocrinol Metab. 2002 Feb;87(2):489-99. doi: 10.1210/jcem.87.2.8182. PMID 11836274
- [Background] Garmendia Madariaga A, Santos Palacios S, Guillen-Grima F, Galofre JC. The incidence and prevalence of thyroid dysfunction in Europe: a meta-analysis. J Clin Endocrinol Metab. 2014 Mar;99(3):923-31. doi: 10.1210/jc.2013-2409. Epub 2014 Jan 1. PMID 24423323
- [Background] Ross DS, Burch HB, Cooper DS, Greenlee MC, Laurberg P, Maia AL, Rivkees SA, Samuels M, Sosa JA, Stan MN, Walter MA. 2016 American Thyroid Association Guidelines for Diagnosis and Management of Hyperthyroidism and Other Causes of Thyrotoxicosis. Thyroid. 2016 Oct;26(10):1343-1421. doi: 10.1089/thy.2016.0229. PMID 27521067
- [Background] Dahl P, Danzi S, Klein I. Thyrotoxic cardiac disease. Curr Heart Fail Rep. 2008 Sep;5(3):170-6. doi: 10.1007/s11897-008-0026-9. PMID 18752767
- [Background] Frost L, Vestergaard P, Mosekilde L. Hyperthyroidism and risk of atrial fibrillation or flutter: a population-based study. Arch Intern Med. 2004 Aug 9-23;164(15):1675-8. doi: 10.1001/archinte.164.15.1675. PMID 15302638
- [Background] Sundaresh V, Brito JP, Wang Z, Prokop LJ, Stan MN, Murad MH, Bahn RS. Comparative effectiveness of therapies for Graves' hyperthyroidism: a systematic review and network meta-analysis. J Clin Endocrinol Metab. 2013 Sep;98(9):3671-7. doi: 10.1210/jc.2013-1954. Epub 2013 Jul 3. PMID 23824415
- [Background] Kaykhaei MA, Shams M, Sadegholvad A, Dabbaghmanesh MH, Omrani GR. Low doses of cholestyramine in the treatment of hyperthyroidism. Endocrine. 2008 Aug-Dec;34(1-3):52-5. doi: 10.1007/s12020-008-9107-5. Epub 2008 Oct 23. PMID 18946743
- [Background] Migneco A, Ojetti V, Testa A, De Lorenzo A, Gentiloni Silveri N. Management of thyrotoxic crisis. Eur Rev Med Pharmacol Sci. 2005 Jan-Feb;9(1):69-74. PMID 15850146
- [Background] Solomon BL, Wartofsky L, Burman KD. Adjunctive cholestyramine therapy for thyrotoxicosis. Clin Endocrinol (Oxf). 1993 Jan;38(1):39-43. doi: 10.1111/j.1365-2265.1993.tb00970.x. PMID 8435884
- [Background] Mercado M, Mendoza-Zubieta V, Bautista-Osorio R, Espinoza-de los Monteros AL. Treatment of hyperthyroidism with a combination of methimazole and cholestyramine. J Clin Endocrinol Metab. 1996 Sep;81(9):3191-3. doi: 10.1210/jcem.81.9.8784067.
- [Background] Jude EB, Dale J, Kumar S, Dodson PM. Treatment of thyrotoxicosis resistant to carbimazole with corticosteroids. Postgrad Med J. 1996 Aug;72(850):489-91. doi: 10.1136/pgmj.72.850.489. PMID 8796215
- [Background] Baeza A, Aguayo J, Barria M, Pineda G. Rapid preoperative preparation in hyperthyroidism. Clin Endocrinol (Oxf). 1991 Nov;35(5):439-42. doi: 10.1111/j.1365-2265.1991.tb03562.x. PMID 1814659
- [Background] Page SR, Sheard CE, Herbert M, Hopton M, Jeffcoate WJ. A comparison of 20 or 40 mg per day of carbimazole in the initial treatment of hyperthyroidism. Clin Endocrinol (Oxf). 1996 Nov;45(5):511-6. doi: 10.1046/j.1365-2265.1996.00800.x. PMID 8977745
- [Background] Ozawa Y, Daida H, Shimizu T, Shishiba Y. Rapid improvement of thyroid function by using glucocorticoid indicated for the preoperative preparation of subtotal thyroidectomy in Graves' disease. Endocrinol Jpn. 1983 Feb;30(1):93-100. doi: 10.1507/endocrj1954.30.93. PMID 6688394
- [Background] Conn HO, Poynard T. Corticosteroids and peptic ulcer: meta-analysis of adverse events during steroid therapy. J Intern Med. 1994 Dec;236(6):619-32. doi: 10.1111/j.1365-2796.1994.tb00855.x. PMID 7989897

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03303053/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03303053/ICF_001.pdf